CLINICAL TRIAL: NCT04034901
Title: Collecte de données Physiologiques en Continu Chez Des Patients en Insuffisance Respiratoire Pendant et après un épisode d'Exacerbation de BPCO
Brief Title: Study of Physiological Signals During and After COPD Exacerbations
Acronym: DACRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosency (Industry)
Collaborators: Slb Pharma (Other); Air de Bretagne (Unknown); Rennes University Hospital (Other); Centre Hospitalier Bretagne Atlantique (Other); Centre Hospitalier de Saint-Malo (Unknown); Centre Hospitalier de Saint-Brieuc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-A00642-55
Record Dates: First submitted 2019-06-28; First posted 2019-07-26 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: COPD; COPD Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring of cardiorespiratory parameters (Experimental): Monitoring of cardiorespiratory parameters with BORA Band
  Interventions: Device: Monitoring of cardiorespiratory parameters with BORA Band

INTERVENTIONS:
Device: Monitoring of cardiorespiratory parameters with BORA Band — The subjects will continuously wear a connected wrist-worn pulse oximeter which will remotely collect the following measurements :
  * Activity
  * Step count
  * Heart rate
  * Respiratory rate
  * Skin temperature
  * SpO2

SUMMARY:
Background : Acute exacerbations of COPD (Chronic Obstructive Pulmonary Disease) are frequent events in the course of the disease and they can deteriorate the respiratory function of the patients, impact their quality of life and even potentially threaten their life. It is therefore crucial to prevent these exacerbations from occurring.

Aim of the study : Investigate how cardiorespiratory parameters of COPD patients differ between exacerbation phases and their nominal state in order to identify predictors of COPD exacerbations.

Study design : Patients admitted at one of the investigation centers on a suspicion of COPD exacerbation will be enrolled on a voluntary basis. Enrolled patients' cardiorespiratory parameters will be monitored with a connected wrist-worn pulse oximeter (BORA Band) during the hospitalisation phase and one month after they have been discharged.

Setting : 4 investigative centers across Brittany

Patients : 50 patients will be enrolled in the study

ELIGIBILITY:
Inclusion Criteria:

* patient known or suspected to suffer from COPD
* patient admitted in pulmonology unit for COPD exacerbation
* patient accepting to use BORA Band during and after hospitalization
* patient accepting to be followed by the partner health care provider for this study (Air de Bretagne)
* patient able to understand French and express their informed consent
* patient affiliated to social security

Exclusion Criteria:

* patient is intubated
* patient already followed by a health care provider other than Air de Bretagne
* investigator assesses that the patient will have difficulties following the protocol
* patient already enrolled in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Variation of heart rate during and after a COPD acute exacerbation | 2 months
  Average heart rate in beats per minute during and after COPD exacerbation will be assessed thanks to a wrist-worn connected pulse oximeter
Variation of respiratory rate during and after a COPD acute exacerbation | 2 months
  Average respiratory rate in cycles per minute during and after COPD exacerbation will be assessed thanks to a wrist-worn connected pulse oximeter
Variation of SpO2 during and after a COPD acute exacerbation | 2 months
  Average SpO2 in percent during and after COPD exacerbation will be assessed thanks to a wrist-worn connected pulse oximeter
Variation of skin temperature during and after a COPD acute exacerbation | 2 months
  Average skin temperature in celcius during and after COPD exacerbation will be assessed thanks to a wrist-worn connected pulse oximeter
Variation of patient activity during and after a COPD acute exacerbation | 2 months
  Average patient activity measured in activity duration per day during and after COPD exacerbation will be assessed thanks to a wrist-worn connected pulse oximeter

SECONDARY OUTCOMES:
Connected wrist-worn pulse oximeter adherence | 2 months
  The mean duration of bora band utilization will be measured (mean number of days and mean number of hours per day)
Patient satisfaction | 2 months
  the patient satisfaction with the connected wrist-worn pulse oximeter will be assessed using a series of yes or no questions about the comfort, the acceptability, the ease of use and the size of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Brinchault, M.D., Principal Investigator — CHU Rennes
Locations (1):
- Chru Pontchaillou, Rennes, France

IPD SHARING:
Plan to Share IPD: No